CLINICAL TRIAL: NCT05012891
Title: Gait Analysis in Patients Undergoing Rehabilitation Due to Lower Extremity Disability or Chronic Pain, Using OneStep Smartphone Application.
Brief Title: Gait Analysis Using OneStep Smartphone Application
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Reuth Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Dana Gefen Doron, Principal Investigator, Reuth Rehabilitation Hospital
Other Study IDs: 0008-20-RRH
Record Dates: First submitted 2020-07-12; First posted 2021-08-19 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain of Left Foot (Finding); Chronic Pain of Right Foot (Finding)
Keywords: Gait analysis; Chronic pain; Smartphone app; Rehabilitation; Adherence and Compliance
MeSH Terms: conditions — Signs and Symptoms; Chronic Pain; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Population: Fifty (n=50) consecutive patients with lower-extremity disability or chronic pain (unilateral or bilateral), undergoing a rehabilitation course in a Day-Care Center setting.
  Interventions: Other: OneStep Smartphone Application

INTERVENTIONS:
Other: OneStep Smartphone Application — OneStep technology is a smartphone application (app) utilizing smartphone sensors to provide ongoing gait diagnostics. The eligible study participants will be asked to download and install the app on their own smartphones and carry the smartphone in their front pants pocket at all times.
  The app will collect the required gait parameters but, will not present them (or any summary thereof) to the study participants or their physiotherapists, in order not to influence the rehabilitation plan.

SUMMARY:
OneStep technology is a smartphone application, utilizing smartphone sensors to provide ongoing gait diagnostics. In this longitudinal study, 50 consecutive patients with lower-extremity disability or chronic pain, will be using the One-Step App, downloaded to their personal smartphones, in parallel with the usual rehabilitation treatments, during a one-month period. Analyzed gait data from the App will be linked with clinical data collected by a team of experts, in order to evaluate the potential use of this App as an objective means to characterize and quantify patients' gait characteristics along the follow-up period, and to objectively assess the patients' adherence and compliance with the rehabilitation regime.

DETAILED DESCRIPTION:
Background:

Patient adherence is a crucial determinant of the rehabilitation process. After injury or surgery, many patients are given specific exercises to conduct unsupervised on their own to aid their recovery. Evidence suggests that noncompliance with the prescribed exercise regime is associated with poor rehabilitation outcomes. OneStep technology is a smartphone application (App), which uses smartphone sensors to provide ongoing gait diagnostics.

Study Objectives:

1. To analyze gait-related parameters collected via the OneStep App in patients with lower extremity disability or chronic pain over a 4-week follow-up period during in-hospital physiotherapy sessions, self-exercises at home, and other daily activities,
2. To objectively assess the patients' adherence and compliance with the prescribed rehabilitation regime. For the purposes of this research, adherence refers to the quantity and frequency of completed home exercises, while compliance refers to the quality of meeting the physiotherapists' walking-related recommendations.
3. To assess gait parameters measured simultaneously on both feet, during standard walking-related tests, (performed under similar conditions on days 1, 14, 28, while using the OneStep App), for between and within-subject comparison.
4. To compare between patients' subjective self-reports on performed physiotherapy workouts at home, the physiotherapists' own subjective assessments on their patients' adherence and compliance, and the objective data collected using the OneStep App

Methods:

Fifty consecutive patients with lower-extremity disability or pain, will be using the One-Step App, downloaded to their personal smartphones, in parallel with the usual rehabilitation treatments, during a one-month period. The study participants will be asked to carry the smartphone with the preinstalled app on them at all times, specifically on their injured foot.

All participants will also be required to undertake standard walking tests at the study initiation day (day 1) and on days 14 and 28 under similar conditions for between and within-subject comparison. Only during these tests will the subjects be using two smartphones preinstalled with the OneStep App, one attached to each leg, for a more accurate gait symmetry assessment.

During these 3 sessions, the study participants, as well as their physiotherapists, will be asked to fill in the study questionnaires.

Hypothesis:

Data collected using the OneStep App will allow an accurate and informative follow-up on patients' adherence and compliance with the rehabilitation regime and assist the physiotherapists in improving the efficacy of the rehabilitation process.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 65 years old.
2. Able to walk independently or with assistance (human/walking aids).
3. Able to speak and read fluently in Hebrew.
4. Admitted for rehabilitation at a rehabilitation hospital day-care center following lower-extremity disability or chronic pain (unilateral or bilateral).
5. Have undergone at least 4 weeks of rehabilitation, but require an additional (at least one month long) rehabilitation course.
6. Subjects must be willing to use their own smartphone device to install the OneStep application for study procedures and to comply with the study protocol.
7. The subjects' smartphone has to be compatible with the OneStep app hardware requirements.

Exclusion Criteria:

1. Subject unable to step on the sore foot.
2. Subject unfit to participate in the study based on the judgment of the study principal investigator.
3. Subjects who are permanently wheelchair-bound.
4. Subjects with known pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a lower-extremity disability or chronic pain (unilateral or bilateral).
  (Chronic pain was defined as pain lasting more than 3 months)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Walking Distance (General Gait Parameter) | One month of follow-up
  The daily walking distance (in meters) as measured by the OneStep App
Walking Time (General Gait Parameter) | One month of follow-up
  The daily walking time (in minutes) as measured by the OneStep App
Step Count (General Gait Parameter) | One month of follow-up
  The daily step count (number of steps) as measured by the OneStep App
Step Time (Leg Specific Parameter) | One month of follow-up
  The average daily step time (in seconds) as measured by the OneStep App
Motion of the Hip Joint (Leg Specific Parameter) | One month of follow-up
  The daily range of hip joint motion (in degrees) as measured by the OneStep App while walking.
Patients' Adherence with the Rehabilitation Regime | One month of follow-up
  The patients' adherence with the rehabilitation regime refers to the quantity and frequency of completed home exercises, converted into an adherence score. Patients' self-reports and physiotherapists' own assessments on patients' adherence will be collected using newly developed questionnaires, while the objective data on patients' adherence will be collected using the OneStep App.
Patients' Compliance with the Rehabilitation Regime | One month of follow-up
  The patients' compliance with the rehabilitation regime refers to the quality of meeting the physiotherapists' walking-related recommendations, converted into a Compliance score. Patients' self-reports and physiotherapists' own assessments on patients' compliance will be collected using newly developed questionnaires, while the objective data on patients' compliance will be collected using the OneStep App.

SECONDARY OUTCOMES:
6-Minute Walk Test (6MWT) | Assessed at days 1, 14 and 28 of the follow-up period
  It is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance (in meters) covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. Each study subject will take this test 3 times: on days 1, 14, and 28 of the follow-up. During these tests, the study participants will be using 2 phones, each preinstalled with the OneStep application and placed on each foot for simultaneous data collection, for within and between-subject comparison.
Timed Up and Go (TUG) Test | Assessed at days 1, 14 and 28 of the follow-up period
  The test measures, in seconds, the time taken by an individual to stand up from a standard armchair walk a distance of 3 meters, turn, walk back to the chair, and sit down again. The subjects are asked to wear their regular footwear and use their customary walking aids. No physical assistance is given. The subjects start the test with their back against the chair, their arms resting on the armrests, and their walking aid at hand. They are instructed that on the word "go" they are to get up and walk at a comfortable and safe pace to a line on the floor 3 meters away, turn, return to the chair and sit down again. Each subject walks through the test once before being timed in order to become familiar with the test. Each subject will take this test 3 times (days 1, 14, and 28). During these tests, the study participants will be using 2 phones, each preinstalled with the OneStep app and placed on each foot for simultaneous data collection, for within and between-subject comparison.
10-Meter Walk Test (10MWT) | Assessed at days 1, 14 and 28 of the follow-up period
  The test is used to measure gait speed (in meters per second) of individuals with gait limitations. A 10-meter straight course will be marked at its beginning and end with tape on the floor. The study participant will be positioned 2 meters behind the first tape line. The subject will then be instructed to walk at a comfortable rate until one passes the second tape line. The timer is started when one crosses the first tape line and stopped when one crosses the second tape line. The 2-meter distances before and after the course serve to minimize the effect of acceleration and deceleration. The test is repeated 3 times and the average time is calculated. Each study subject will take these tests on 3 occasions (days 1, 14, and 28). During these tests, the study participants will be using 2 phones, each preinstalled with the OneStep application and placed on each foot for simultaneous data collection, for within and between-subject comparison.

OTHER OUTCOMES:
Brief Pain Inventory (BPI) | Assessed at days 1, 14 and 28 of the follow-up period
  The Brief Pain Inventory (BPI) is a multidimensional measurement tool, which contains a figure of the body on which patients can mark their painful sites. The 4-item BPI Pain Severity Subscale is used to measure overall pain: at its worst, at its least, on average (all - over the last 24 hours) and at present, using a 0-10 numeric rating scale, where 0 indicates no pain and 10 corresponds to "severe or excruciating pain as bad as you can imagine". The BPI has seven Numeric Rating Scales (NRS) that show how the pain interferes with function, mood, and enjoyment.
Lower Extremity Functional Scale (LEFS) | Assessed at days 1, 14 and 28 of the follow-up period
  The LEFS is a 20-item self-report measure of physical function. Each item is rated on a five-point scale (0-4), with lower scores representing greater difficulty. Total scores can range from 0 to 80. Function is defined as follows: extreme difficulty or unable to perform activity (0-19 points), quite a bit of difficulty (20-39 points), moderate difficulty (40-59 points), a little bit of difficulty (60-79 points), and no difficulty (80 points).
ABC Confidence Scale | Assessed at days 1 and 28 of the follow-up period
  Self administered 16 question assessment in which subjects are instructed to answer each question with a percentage of confidence that they will not fall while performing a given task from 0%-100%, with 0% being "not confident" and 100% being "confident". Scores 80% or higher indicate a high level of physical functioning, 50-80% indicate a moderate level of physical functioning and scores less than 50% indicate a low level of physical functioning.
Video Documentation | Recorded on days 1, 14 and 28 of the follow-up period
  Subjects will be videotaped during their performance in the Six Minute Walk Test, Ten Meter Walk Test and Timed Up and Go Test to visually assess and document any changes in gait parameters, from baseline measurements. The videotaping procedures will focus only on the subject's lower extremities.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Gefen Doron, MD, Principal Investigator — Reuth Rehabilitation Hospital
Locations (1):
- Reuth Rehabilitation Hospital, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided